CLINICAL TRIAL: NCT02473029
Title: Interest of Medical Imaging in the Diagnostic Strategy Vis a Vis a Suspected Horton Disease
Acronym: HORTIM
Status: Terminated | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: GEL_2014_01
Record Dates: First submitted 2015-06-12; First posted 2015-06-16 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Horton Disease
MeSH Terms: conditions — Giant Cell Arteritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cases: Patients admitted to a tertiary hospital, with a clinical suspicion of Horton disease
  Interventions: Radiation: Vascular tomodensitometry; Other: Magnetic resonance angiography; Other: Vascular ultrasonography; Other: Retinal angiography; Other: Retinal optical coherence tomography

INTERVENTIONS:
Radiation: Vascular tomodensitometry
Other: Magnetic resonance angiography
Other: Vascular ultrasonography
Other: Retinal angiography
Other: Retinal optical coherence tomography

SUMMARY:
The study aims at measuring the sensitivity and specificity of a series of imaging signs (recorded by magnetic resonance angiography, vascular tomodensitometry, vascular ultrasonography, retina angiography and retina optic coherence tomography) for the diagnosis of Horton disease, the gold standard being the result of temporal artery biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the Fondation Ophtalmologique Adolphe de Rothschild and suspected to suffer from Horton disease, based on the presence of 3 or more major criteria, or 2 major criteria and at least one minor criteria.

Major criteria : Age > 50 ans ; headache ; intermittent jaw or tongue pain ; visual impairment ; ESR > 50 mm at 1h and/or CRP > 8mg/l.

Minor criteria: temporal artery or scalp tenderness ; facial pain or tenderness ; fever >38°C, weight loss >10%, anorexia, fatigue.

Exclusion Criteria:

* Autoimmune disease
* Active infectious condition
* Malignant disease
* Condition counterindicating one or several of the protocol's imaging procedures : allergy to iodine and/or renal insufficiency and/or claustrophobia and/or metallic foreign body...

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Fondation Ophtalmologique Adolphe de Rothschild with a suspected Horton disease
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
MRI angiography mural inflammation | Baseline
  Presence of signs of artery mural inflammation in T1 sequence of MRI angiography

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique A. de Rotchschild, Paris, France